CLINICAL TRIAL: NCT06030752
Title: Washed Microbiota Transplantation (WMT) for Autism Spectrum Disorder (ASD)
Brief Title: WMT for Autism Spectrum Disorder (ASD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WMT-ASD-2023
Record Dates: First submitted 2023-05-25; First posted 2023-09-11 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder
Keywords: fecal Microbiota Transplantation; Autism spectrum disorder; Gut microbiota; Gut-brain axis
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Washed microbiota transplantation (Experimental): WMT
  Interventions: Drug: Washed Microbiota Transplantation

INTERVENTIONS:
Drug: Washed Microbiota Transplantation — The prepared microbiota suspension was infused into the participates' lower gut.
  Other Names: Fecal Microbiota Transplantation

SUMMARY:
Autism Spectrum Disorder (ASD) is a group of serious neurodevelopmental disorders. A significant comorbidity exists between ADHD and ASD: 30%-50% of individuals with ASD exhibit ADHD symptoms, and two-thirds with ADHD show ASD traits. Intestinal microbial disturbance is common in children with ASD. A great deal of evidence shows that intestinal microbes can influence the brain to play its role through "gut-brain-microbiota axis". We intend to explore the role of Washed Microbiota Transplantation in improving symptoms of children in ASD with or without ADHD; To study the potential etiological mechanism of WMT for the neurodevelopmental disorders.

DETAILED DESCRIPTION:
Very few literatures reported the clinical use of microbiota or bacteria for Autism Spectrum Disorder. The most effective strategy for reconstruction of gut microbiota should be fecal microbiota transplantation (WMT). Washed microbiota transplantation (WMT) can significantly reduce FMT-related AEs by removing parasite eggs, fecal particles, and fungi through a series of automated washing procedures. This study aims to evaluate the efficacy and safety of FMT for ASD. Patients received repeated WMT with fecal from healthy donors. Microbiota analysis will also be performed on both the donor and recipient stool sample prior to transplantation, and on the recipient sample at 3 month post transplantation. This study sought to evaluate the efficacy of washed microbiota transplantation (WMT) in children with ASD and explore the role of washed bacteria transplantation in improving ASD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with an established diagnosis of ADHD or ADHD + ASD according to the Diagnostic and Statistical Manual Of Mental Disorders Fifth Edition;.
* Age 3-17 years.
* Received stable treatments for ≥1 month preceding WMT

Exclusion Criteria:

* Their guardian could not understand the questionnaires or provide informed consent.
* Diagnosed with a single-gene disorder, major brain malformations, gastrointestinal diseases (ulcerative colitis, Crohn's disease, or eosinophilic esophagitis)
* Had severe comorbidities including cardiopulmonary failure, severe liver, and kidney diseases, severe infection, tumors, etc.
* Accompanied with other life-threatening disorders required emergency treatment.
* Unable to tolerate colonoscopy or anesthesia.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2027-04-04 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the Autism Behavior Checklist (ABC) in ASD children | baseline, 1 month , 3 months, 6 months post transplantation
  ABC is a scale used for nonadaptive behaviors created to screen and indicate the probability of a diagnosis of autism. The questionnaire including 57 items related to five areas: sensorial, relational, use of body and objects, and social skills. Scale score> 67 strongly suggests the presence of autism.
Change in Autism Treatment Evaluation Checklist (ATEC) in ASD children | baseline, 1 month,3 months, 6 months post transplantation
  ASD symptoms will be assessed using the Chinese version of the Autism Treatment Evaluation Checklist (ATEC), which comprise four subscales to measure child speech/language/communication, sociability, sensory/cognitive awareness, and health/physical/behavior. The scale has 77 items that are scored by parents. The health/physical/behavior subscale is rated using a 0 (not a problem)-to-3 (serious problem) point scale, whereas the other three subscales are rated using a 0 (not true)-to-2 (very true) point scale. Higher scores represent more ASD symptoms.

SECONDARY OUTCOMES:
Evaluate the difference of the gut microbe composition between children with ASD and healthy children by sequencing faecal metagenome. | Fecal samples from ASD and healthy children were collected at baseline and 3 month, 6 months post transplantation.
  The composition of the gut microbe was evaluated by sequencing faecal metagenome. We evaluate the differences in the structure of the flora and its metabolism between the two at the phylum, genus and species levels of the intestinal flora and control children, and to develop a model for predicting the structure of the flora.
The Sleep Disturbance Scale for Children | baseline, 1 month, 3 months, 6 months post transplantation
  The Sleep Disturbance Scale for Children (SDSC) was used to assess sleep quality in children with ASD. It had 26 items, each with a score from 0-4. Higher SDSC scores indicated poorer sleep quality
The Gastrointestinal Symptom Rating Scale | baseline, 1 month, 3 months, 6 months post transplantation
  The Gastrointestinal Symptom Rating Scale (GSRS) was used to assess gastrointestinal symptoms. It was a 7-point Likert scale questionnaire with 15 items. The 15 items can be divided into 5 dimensions: abdominal pain (3 items), reﬂux (2 items), dyspepsia (4 items), diarrhea (3 items), and constipation (3 items).
Clinical Global Impressions-Improvement | baseline, 1 months, 3 months, 6 months post transplantation
  The Clinical Global Impressions-Improvement (CGI-I) evaluated by experienced clinician was used to assess the symptom changes relative to baseline, rated on a 7-point scale from 1 (very much improved) to 7 (very much worse) [26]. CGI-I = 1 or 2 was considered a clinical response.
The Chinese version of Swanson, Nolan, and Pelham-IV (SNAP-IV) | At baseline, 1 month, 3 months and 6 months after WMT
  It was a 26-item questionnaire that measured three of the ADHD symptoms, inattention (items 1-9), hyperactivity (items 10-18), and oppositional defiant disorder (items 19-26). The 26-item checklist was scored on a 4-point Likert scale ranging between Not At All (0) and Very Much (3).
Conners' Parent Rating Scale-Revised (CPRS-R) | At baseline, 1 month, 3 months and 6 months after WMT
  The CPRS-R was composed of 10 items derived from the Revised Conners Parent Rating Scale. It used a 4-point Likert scale (range: 0-30), with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (2):
- China (2):
  - Department of Microbiota Medicine & Medical Centre for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - SIR RUN RUN hospital of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirota T, King BH. Autism Spectrum Disorder: A Review. JAMA. 2023 Jan 10;329(2):157-168. doi: 10.1001/jama.2022.23661. PMID 36625807
- [Background] Solmi M, Radua J, Olivola M, Croce E, Soardo L, Salazar de Pablo G, Il Shin J, Kirkbride JB, Jones P, Kim JH, Kim JY, Carvalho AF, Seeman MV, Correll CU, Fusar-Poli P. Age at onset of mental disorders worldwide: large-scale meta-analysis of 192 epidemiological studies. Mol Psychiatry. 2022 Jan;27(1):281-295. doi: 10.1038/s41380-021-01161-7. Epub 2021 Jun 2. PMID 34079068
- [Background] Brugha TS, Spiers N, Bankart J, Cooper SA, McManus S, Scott FJ, Smith J, Tyrer F. Epidemiology of autism in adults across age groups and ability levels. Br J Psychiatry. 2016 Dec;209(6):498-503. doi: 10.1192/bjp.bp.115.174649. Epub 2016 Jul 7. PMID 27388569
- [Background] Khachadourian V, Mahjani B, Sandin S, Kolevzon A, Buxbaum JD, Reichenberg A, Janecka M. Comorbidities in autism spectrum disorder and their etiologies. Transl Psychiatry. 2023 Feb 25;13(1):71. doi: 10.1038/s41398-023-02374-w. PMID 36841830
- [Background] Liang X, Haegele JA, Tse AC, Li M, Zhang H, Zhao S, Li SX. The impact of the physical activity intervention on sleep in children and adolescents with autism spectrum disorder: A systematic review and meta-analysis. Sleep Med Rev. 2024 Apr;74:101913. doi: 10.1016/j.smrv.2024.101913. Epub 2024 Feb 23. PMID 38442500
- [Background] Chen Y, Fang H, Li C, Wu G, Xu T, Yang X, Zhao L, Ke X, Zhang C. Gut Bacteria Shared by Children and Their Mothers Associate with Developmental Level and Social Deficits in Autism Spectrum Disorder. mSphere. 2020 Dec 2;5(6):e01044-20. doi: 10.1128/mSphere.01044-20. PMID 33268567
- [Background] Jacob S, Veenstra-VanderWeele J, Murphy D, McCracken J, Smith J, Sanders K, Meyenberg C, Wiese T, Deol-Bhullar G, Wandel C, Ashford E, Anagnostou E. Efficacy and safety of balovaptan for socialisation and communication difficulties in autistic adults in North America and Europe: a phase 3, randomised, placebo-controlled trial. Lancet Psychiatry. 2022 Mar;9(3):199-210. doi: 10.1016/S2215-0366(21)00429-6. Epub 2022 Feb 10. PMID 35151410
- [Background] Hung LY, Margolis KG. Autism spectrum disorders and the gastrointestinal tract: insights into mechanisms and clinical relevance. Nat Rev Gastroenterol Hepatol. 2024 Mar;21(3):142-163. doi: 10.1038/s41575-023-00857-1. Epub 2023 Dec 19. PMID 38114585
- [Background] Liu NH, Liu HQ, Zheng JY, Zhu ML, Wu LH, Pan HF, He XX. Fresh Washed Microbiota Transplantation Alters Gut Microbiota Metabolites to Ameliorate Sleeping Disorder Symptom of Autistic Children. J Microbiol. 2023 Aug;61(8):741-753. doi: 10.1007/s12275-023-00069-x. Epub 2023 Sep 4. PMID 37665552
- [Background] Wan Y, Zuo T, Xu Z, Zhang F, Zhan H, Chan D, Leung TF, Yeoh YK, Chan FKL, Chan R, Ng SC. Underdevelopment of the gut microbiota and bacteria species as non-invasive markers of prediction in children with autism spectrum disorder. Gut. 2022 May;71(5):910-918. doi: 10.1136/gutjnl-2020-324015. Epub 2021 Jul 26. PMID 34312160
- [Background] Zhang T, Lu G, Zhao Z, Liu Y, Shen Q, Li P, Chen Y, Yin H, Wang H, Marcella C, Cui B, Cheng L, Ji G, Zhang F. Washed microbiota transplantation vs. manual fecal microbiota transplantation: clinical findings, animal studies and in vitro screening. Protein Cell. 2020 Apr;11(4):251-266. doi: 10.1007/s13238-019-00684-8. Epub 2020 Jan 9. PMID 31919742
- [Background] Nanjing consensus on methodology of washed microbiota transplantation. Chin Med J (Engl). 2020 Oct 5;133(19):2330-2332. doi: 10.1097/CM9.0000000000000954. No abstract available. PMID 32701590